CLINICAL TRIAL: NCT06004284
Title: Effect of Exercise Given to Factory Workers With Ergonomics Training on Pain and Functionality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, assistant professor, Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uskudar69
Record Dates: First submitted 2023-08-09; First posted 2023-08-22 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Work-related Illness; Work Accident; Occupational Diseases
Keywords: Workers; pain; exercise; ergonomics; Functionality
MeSH Terms: conditions — Occupational Diseases; Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be given exercise practices along with ergonomics training.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Active Comparator): Only ergonomics training will be given to the control group.
  Interventions: Other: control
- exercise group (Experimental): Participants will be given training including stretching and core exercises along with ergonomics training.
  Interventions: Other: exercise group

INTERVENTIONS:
Other: control — Ergonomics training will be given to each of the control group participants individually. The content of this training will include "what is ergonomics, the purpose of ergonomics, musculoskeletal diseases in employees, work-related musculoskeletal risk fa
  Arms: control group
Other: exercise group — The exercise training program will be applied for 8 weeks, 3 days a week and for an average of 20-30 minutes. After the maneuver is taught, stretching exercises lasting 5 minutes for warm-up purposes and posture and core exercises lasting 25 minutes will be taught. Among the stretching exercises, quadratus lumborum stretching, hamstring stretching, erector spina stretching, hip extensor stretching exercises will be applied. Posterior pelvic tilt exercise will be performed as a control and smoothing exercise for the vertebrae of the lumbar and pelvic region. Among the core stabilization exercises, bridging, plank, plank in side lying, abdominal strengthening, cross arm leg lifting exercises in crawling position will be performed. Each exercise position will be required to be maintained for 8 seconds and to do 10-15 repetitions.
  Arms: exercise group

SUMMARY:
The aim of this study is to evaluate the effects of ergonomics training with exercises applied on factory workers with low back pain on pain, functionality, sleep and fatigue.

DETAILED DESCRIPTION:
The study was planned as a randomized controlled trial. Workers between the ages of 18 and 60 working in a plastic casting factory in Gebze/Kocaeli with back and low back pain will be included in the study. Participants will be divided into two groups using a simple randomization method. Ergonomics training will be given to the first group together with core stabilization exercises; The second group will be given only ergonomics training. The exercises they will do will be explained to the participants individually and will be supported by an exercise brochure. Participants will be asked to do the given exercises 3 days a week and continue for 8 weeks. Follow-up of the given exercises will be done with the exercise follow-up chart. Persons with psychological or physical disabilities who can exercise regularly will not be included in the study. In order to collect data on the sociodemographic characteristics of the participants, a personal information form will be prepared by the researcher and the participants will be asked to fill in this form. In order to collect data from the participants; "McGill Pain Questionnaire (Short)" and "Visual Analog Scale" to collect information on pain; "Fatigue Severity Scale" will be used to determine fatigue levels, "Pittsburgh Sleep Quality Questionnaire" will be used to determine sleep quality, and "Oswestry Low Back Pain Scale" will be used to evaluate functionality. The questionnaires will be repeated before and after the study. The data before and after the intervention will be analyzed statistically.

ELIGIBILITY:
Inclusion Criteria:

* be between the ages of 18-65,
* Having low back pain in the last 3 months
* Visual Pain Scale (VAS) >4
* No surgical intervention in the last 6 months,

Exclusion Criteria:

* Not being cooperative desk work
* Presence of psychological problems,
* Using sleeping pills
* Presence of neurological and orthopedic disease.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

PRIMARY OUTCOMES:
The McGill Pain Questionnaire (MPQ) | 10 weeks
  McGill pain questionnaire-short form is used to evaluate patients' pain in terms of feeling and sensory. Pain level is defined with 15 words consisting of 11 sensory and 4 affective words. From these descriptive words, the patient should choose an answer that is compatible with him/her as "no (0)", "mild (1)", "moderate (2)", "severe (3)". In addition, the pain felt during the survey is measured with the VAS, and the total pain intensity of the pain is measured with a 6-point Likert scale. Pain is defined as "absent (0)" and "unbearable (5)" on the Likert scale. In total, pain scores between 0-45 (no pain=0, severe pain=45).
Oswestry Low Back Pain Disability Questionnaire | 10 weeks
  It was developed to measure the functionality of individuals. The scale determines functional disability for activities such as sitting, walking, personal care, lifting, social life, travel, and sleep. There are 10 questions in this scale. Each question has 6 options. Participants are asked to choose the definition that best describes their situation from these options. A score of 0-5 is assigned for each of the sentences, and the highest possible score is 50 points. It is evaluated as mild between 1 and 10 points, moderate between 11 and 30 points, and severe between 31 and 50 points.
Fatigue Severity Scale (FSS) | 10 weeks
  This scale consists of 9 questions and each option has a score between 0-7. A score of 0 is expressed as "strongly disagree", while a score of 7 is expressed as "agree". The maximum score is 7, and it is recorded that people have a significant degree of fatigue for 4 points and above.
The Pittsburgh Sleep Quality Index (PSQI) | 10 weeks
  Pittsburgh Sleep Quality Index; It evaluates sleep duration, sleep disturbance, sleep efficiency, subjective sleep quality, sleep medication use, daytime dysfunction, and sleep delay and consists of a total of 24 questions. 19 of them are self-report scales and 5 of them consist of questions to be answered by a friend or spouse. There are 7 components with 18 questions scored in the scale, and each component is evaluated between 0 and 3 points. The total score ranges from 0 to 21, and 5 or more is an indicator of "poor sleep quality".

CONTACTS AND LOCATIONS:
Overall Officials: Elif PEHLEVAN, Study Chair — Uskudar University
Locations (1):
- Üsküdar Unıversıty, Gebze, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Erick PN, Smith DR. A systematic review of musculoskeletal disorders among school teachers. BMC Musculoskelet Disord. 2011 Nov 17;12:260. doi: 10.1186/1471-2474-12-260. PMID 22087739
- [Background] Bell JA, Burnett A. Exercise for the primary, secondary and tertiary prevention of low back pain in the workplace: a systematic review. J Occup Rehabil. 2009 Mar;19(1):8-24. doi: 10.1007/s10926-009-9164-5. Epub 2009 Feb 14. PMID 19219537
- [Background] Biman S, Maharana S, Metri KG, Nagaratna R. Effects of yoga on stress, fatigue, musculoskeletal pain, and the quality of life among employees of diamond industry: A new approach in employee wellness. Work. 2021;70(2):521-529. doi: 10.3233/WOR-213589. PMID 34633352
- [Background] Coulombe BJ, Games KE, Neil ER, Eberman LE. Core Stability Exercise Versus General Exercise for Chronic Low Back Pain. J Athl Train. 2017 Jan;52(1):71-72. doi: 10.4085/1062-6050-51.11.16. Epub 2016 Nov 16. PMID 27849389
- [Background] Abdollahi T, Pedram Razi S, Pahlevan D, Yekaninejad MS, Amaniyan S, Leibold Sieloff C, Vaismoradi M. Effect of an Ergonomics Educational Program on Musculoskeletal Disorders in Nursing Staff Working in the Operating Room: A Quasi-Randomized Controlled Clinical Trial. Int J Environ Res Public Health. 2020 Oct 8;17(19):7333. doi: 10.3390/ijerph17197333. PMID 33049927
- [Background] Jaromi M, Nemeth A, Kranicz J, Laczko T, Betlehem J. Treatment and ergonomics training of work-related lower back pain and body posture problems for nurses. J Clin Nurs. 2012 Jun;21(11-12):1776-84. doi: 10.1111/j.1365-2702.2012.04089.x. PMID 22594388